CLINICAL TRIAL: NCT00038779
Title: Megadose T-cell Depleted HLA-nonidentical Blood Progenitor Cell Transplantation for Patients With Hematologic Malignancies or Bone Marrow Failure States
Brief Title: Blood Transplantation for Patients With Hematologic Malignancies or Bone Marrow Failure States
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM96-122
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Leukemia; Non Hodgkin's Lymphoma; Aplastic Anemia
Keywords: Lymphoma; CML; CLL; AML; ALL; MDS; AA
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin; Anemia, Aplastic; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Megadose T cell depleted (Experimental)
  Interventions: Procedure: Megadose T-cell Depleted HLA-nonidentical Blood Progenitor Cell Transplantation

INTERVENTIONS:
Procedure: Megadose T-cell Depleted HLA-nonidentical Blood Progenitor Cell Transplantation

SUMMARY:
The purpose of this study is to assess early treatment failure within 100 days and to assess the effect of this regimen on engraftment, GVHD, immune recovery, relapse of malignancy and survival.

ELIGIBILITY:
* Patients with acute leukemia, lymphoma that failed to respond or relapsed after chemotherapy or CML beyond first chronic phase.
* Patients with aplastic anemia or myelodysplasia which failed to respond to primary therapy are eligible.
* Patients with low grade lymphoma or CLL will only be eligible if they failed two chemotherapy regimens and have stage IV disease.
* Patients must be <age 50 with a related haploidentical donor (phenotypically one, two or three HLA A, B and DR antigen mismatched) donor.
* Patients should have adequate hepatic and renal function with a bilirubin of less than or equal to 1.5mg%, SGPT less than or equal to 3x the upper limits of normal, and creatine less than or equal to 1.5mg%.
* Patients with serious intercurrent medical illness are not eligible.
* Patients and their donors must provide written informed consent.

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 1996-08-14 (Actual); Primary Completion 2004-09-20 (Actual); Study Completion 2004-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States